CLINICAL TRIAL: NCT07100366
Title: Comparing Sarcopenia, Physical, Psychological and Social Frailty in Hospitalized Older Women Congestive Heart Failure (CHF) in Metropolitan and Rural Settings: a 3-Year Longitudinal Study Incorporating Information and Communication Technology (ICT) Interventions.
Brief Title: Comparing Sarcopenia , Physical, Psychological and Social Frailty in Hospitalized Older Women Congestive Heart Failure in Metropolitan and Rural Settings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202500795B0
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: 65 Years Older; CHF - Congestive Heart Failure; Social Communication; Sarcopenia in Elderly
Keywords: Frailty; Sarcopenia; Social Frailty; Congestive Heart Failure; Older Women; ICT Intervention; Metropolitan; Rural
MeSH Terms: conditions — Heart Failure; Communication; Frailty; Sarcopenia | interventions — Community Psychiatry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention)
- ChatGPT intervention (Experimental): ChatGPT intervention
  Interventions: Behavioral: ChatGPT
- Community social participation group (Experimental)
  Interventions: Behavioral: community social

INTERVENTIONS:
Behavioral: ChatGPT — Phase 3:In Experimental Group 1, participants will be invited to use the ICT app, which they are encouraged to engage with for at least 15 minutes daily. This app is designed to actively monitor the users' emotional status and automatically notify both the research team and family members if any negative mood is detected.
  Arms: ChatGPT intervention
Behavioral: community social — Phase 3:In Experimental Group 2, participants will be encouraged to increase their social participation through community-based activities, while the Control Group will continue with their routine lifestyle.
  Arms: Community social participation group

SUMMARY:
Frailty-encompassing sarcopenia, physical, psychological, and social frailty-is common among older adults with congestive heart failure (CHF) and contributes to adverse outcomes such as rehospitalization, mortality, and poor quality of life. However, few studies have compared these conditions in congestive heart failure (CHF) patients, particularly in elderly women in Taiwan, and effective, tailored Information and Communication Technology (ICT) interventions are scarce.

This three-year study aims to (1) compare baseline characteristics and incidence rates of sarcopenia, physical, psychological, and social frailty among hospitalized older women with congestive heart failure (CHF) in metropolitan versus rural hospitals; (2) evaluate risk factors associated with physical, psychological, and social frailty; (3) monitor health outcomes (rehospitalization, mortality, quality of life) during a one-year follow-up; and (4) assess the effectiveness of an Information and Communication Technology (ICT) intervention designed to enhance social connectivity and emotional well-being.

In Phase 1, clinical data-including ejection fraction, congestive heart failure (CHF) stage, and comorbidity -will be collected using the 2024 Guidelines of the Taiwan Society of Cardiology, while sarcopenia will be identified via Asian Working Group for Sarcopenia (AWGS) guidelines. Physical, psychological, and social frail will be measured with the Tilburg Frailty Indicator (TFI) and Makizako's Social Frailty Questionnaire, respectively, and physical activity will be assessed using the IPAQ-S.

Phase 2 will involve quarterly follow-ups over one year to compare health outcomes between metropolitan and rural settings, and to develop a predictive model of these outcomes. Phase 3 employs a quasi-experimental design with 90 participants randomized into three groups: an Information and Communication Technology (ICT) intervention group (using a dedicated app for at least 15 minutes daily, which monitors emotional status), a community-based social participation group, and a control group maintaining routine care. Key outcomes (mood, physical activity, frailty measures, and clinical status) will be assessed at baseline, immediately post-intervention, and three months thereafter.

This study is expected to identify significant differences between settings and demonstrate that a tailored Information and Communication Technology (ICT) intervention can improve social connectivity and clinical outcomes in older women with congestive heart failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 65 years or older.
* Diagnosis of CHF with a left ventricular ejection fraction (EF) of less than 40%
* Ability to communicate effectively in Mandarin or Taiwanese.

Exclusion Criteria:

* Patients diagnosed with unstable heart failure
* Severe Comorbidities, conditions such as end-stage renal disease, advanced hepatic dysfunction, or terminal malignancies.
* Severe cognitive deficits that impede the ability to provide informed consent or participate in study interventions.
* Uncorrected visual or hearing impairments that would hinder effective communication or interaction with the ChatGPT application.
* Active psychiatric conditions, including major depression or psychosis, that could interfere with study participation or adherence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Tilburg Frailty Indicator (TFI) | Baseline, 3-month follow-up
  Assesses multidimensional frailty across physical, psychological, and social domains using a 15-item questionnaire. It consists of two parts: the first part gathers data on determinants of frailty (e.g., age, gender, marital status), while the second part includes 15 items divided into physical (8 items), psychological (4 items), and social (3 items) domains. This instrument offers a holistic view of an individual's frailty status. The TFI has shown good internal consistency (Cronbach's α = 0.79) and predictive validity for adverse outcomes, including functional decline and mortality.
  Score range : 0-15 Scores 0-4 Scores: non-frail ; 5 Scores or more: frail
Makizako Social Frailty Index | Baseline, 3-month follow-up
  Assesses social frailty through a set of 5 questions related to social participation, activities, and support networks. The questionnaire has demonstrated good test-retest reliability and criterion validity in predicting adverse health outcomes such as reduced physical activity and functional decline. These instruments collectively provide a comprehensive framework for assessing physical, psychological, and social frailty, especially in studies involving older adults.
  Score range : 0-5 Scores 0 Scores: non-Social Frailty ;
  1. Scores : Pre-Social Frailty ;
  2. Scores or more: Social Frailty
International Physical Activity Questionnaire - Short Form (IPAQ-S) | Baseline, 3-month follow-up
  A self-reported measure assessing physical activity over the last seven days. It categorizes activity levels based on frequency and intensity, covering domains such as walking, moderate activity, and vigorous activity.
  Calculate MET-minutes/week Category 1: Low No activity is reported & Activity does not meet the criteria for Moderate or High categories.
  Category 2: Moderate
  Meets any of the following:
  3 or more days of vigorous activity of at least 20 min/day ; 5 or more days of moderate activity and/or walking of at least 30 min/day ; 5 or more days of any combination of walking, moderate, or vigorous activities, achieving at least 600 MET-min/week Category 3: Vigorous
  Meets either of the following:
  At least 3 days, accumulating at least 1500 MET-min/week, OR 7 or more days of any combination of activities totaling ≥3000 MET-min/week
Minnesota Living with Heart Failure Questionnaire（MLHFQ） | Baseline, 3-month follow-up
  One of the most widely used health-related quality of life questionnaires for patients with CHF.
  Score range : 0-105 Scores 0-24 Scores: Low impact of heart failure on life ; 25-45 Scores: Moderate impact of heart failure on life ; 46 Scores or more: Serious impact of heart failure on life
UCLA Loneliness Scale | Baseline, 3-month follow-up
  Measures subjective feelings of loneliness and social isolation. Score range : 6-18 Scores ; Higher total scores indicate greater feelings of loneliness.
Geriatric Depression Scale (GDS-15) | Baseline, 3-month follow-up
  A shorter 15-item version and designed to screen for depression in older adults.
  Each depressive answer scores 1 point. Some items count "Yes" as a point. Some items count "No" as a point. The maximum total score is 15. Items Scored as 1 Point for a "Yes" Answer:1, 5, 7, 11, 13 Items Scored as 1 Point for a "No" Answer:2, 3, 4, 6, 8, 9, 10, 12, 14, 15 Interpretation of Scores 0-6: Normal (no depression) ; 7-10: Moderate depression ; 11-15: Severe depression
Clinical Frailty Scale (CFS) | Baseline, 3-month follow-up
  A 9-point scale that evaluates an individual's level of frailty based on their physical functioning and overall health status.
  Scoring Range The scale ranges from 1 to 9, with higher scores indicating greater frailty.

IPD SHARING:
Plan to Share IPD: No